CLINICAL TRIAL: NCT03926338
Title: Neoadjuvant PD-1 Blockade by Toripalimab With or Without Celecoxib in Mismatch-repair Deficient or Microsatellite Instability-high Locally Advanced Colorectal Cancer (PICC)
Brief Title: Neoadjuvant Toripalimab With or Without Celecoxib in dMMR/MSI-H Colorectal Cancer
Acronym: PICC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: GIHSYSU-14
Record Dates: First submitted 2019-04-20; First posted 2019-04-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Mismatch Repair-deficient (dMMR); Microsatellite Instability-high (MSI-H); Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — Celecoxib; toripalimab; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: The PICC trial is an investigator-initiated, multi-cohort platform trial designed to evaluate the efficacy and safety of neoadjuvant toripalimab, with or without celecoxib, in patients with mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) locally advanced colorectal cancer. Each cohort within the PICC platform was independently conducted and analyzed according to prespecified objectives.
Who Masked: Outcomes Assessor
Masking Description: Patients and treating physicians are not masked to the study treatment. Investigators who assess radiological, endoscopic, and pathological responses are masked to the treatment allocation and to all other study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PICC-1 exploratory cohort (Experimental): Neoadjuvant toripalimab with or without celecoxib for 6 cycles
  Interventions: Drug: Neoadjuvant toripalimab plus celecoxib for 6 cycles; Drug: Neoadjuvant toripalimab monotherapy for 6 cycles
- PICC-2 cohort (Experimental): Neoadjuvant toripalimab with or without celecoxib for 12 cycles
  Interventions: Drug: Neoadjuvant toripalimab plus celecoxib for 12 cycles; Drug: Neoadjuvant toripalimab monotherapy for 12 cycles
- PICC-3 cohort (Experimental): Toripalimab plus celecoxib as neoadjuvant or definitive therapy
  Interventions: Drug: Toripalimab plus celecoxib as neoadjuvant or definitive therapy

INTERVENTIONS:
Drug: Neoadjuvant toripalimab plus celecoxib for 6 cycles — Toripalimab was administered intravenously over 30 minutes at a dose of 3 mg per kilogram on day 1 of each 14-day cycle, every 2 weeks for a total of 6 cycles, and celecoxib was given orally at 200 mg twice daily from day 1 to day 14 of each cycle, followed by surgery.
  Other Names: Toripalimab; Celecoxib
  Arms: PICC-1 exploratory cohort
Drug: Neoadjuvant toripalimab monotherapy for 6 cycles — Toripalimab was administered intravenously over 30 minutes at a dose of 3 mg per kilogram on day 1 of each 14-day cycle, every 2 weeks for a total of 6 cycles, followed by surgery.
  Other Names: Toripalimab
  Arms: PICC-1 exploratory cohort
Drug: Neoadjuvant toripalimab plus celecoxib for 12 cycles — Toripalimab was administered intravenously over 30 minutes at a dose of 3 mg per kilogram on day 1 of each 14-day cycle, every 2 weeks for a total of 12 cycles, and celecoxib was given orally at 200 mg twice daily from day 1 to day 14 of each cycle, followed by surgery.
  Other Names: Toripalimab; Celecoxib
  Arms: PICC-2 cohort
Drug: Neoadjuvant toripalimab monotherapy for 12 cycles — Toripalimab was administered intravenously over 30 minutes at a dose of 3 mg per kilogram on day 1 of each 14-day cycle, every 2 weeks for a total of 12 cycles, followed by surgery.
  Other Names: Toripalimab
  Arms: PICC-2 cohort
Drug: Toripalimab plus celecoxib as neoadjuvant or definitive therapy — Toripalimab was administered intravenously over 30 minutes at a dose of 3 mg per kilogram on day 1 of each 14-day cycle, every 2 weeks for a total of 12 cycles, and celecoxib was given orally at 200 mg twice daily from day 1 to day 14 of each cycle, followed by surgery or non-operative management based on restaging (non-operative management was recommended for patients with a complete clinical response).
  Other Names: Toripalimab; Celecoxib
  Arms: PICC-3 cohort

SUMMARY:
Colorectal cancer of Mismatch Repair-deficient (dMMR)/ Microsatellite Instability-high (MSI-H) accounts for approximately 15% of all colorectal cancer patients, with a higher proportion in right colon cancer. Previous studies have found that colon cancer patients with dMMR/MSI-H cannot benefit from 5-fluorouracil (5-FU) adjuvant chemotherapy. Once patients have distant metastases, they are not sensitive to traditional palliative chemotherapy, and the prognosis is significantly worse than that of mismatch repair-proficient (pMMR)/microsatellite stability (MSS). A phase II clinical study of anti-PD-1 immunotherapy based on mismatch repair (MMR) status published in 《N Engl J Med》 showed that the objective response rate (ORR) of advanced colorectal cancer patients with dMMR received anti-PD-1 is 40%, and a longer response time can be obtained compared to conventional chemotherapy.

Anti-PD-1 neoadjuvant therapy has proven to be safe and feasible in lung cancer, bladder cancer and malignant melanoma, and can achieve more than 40% of major pathological response. However, there are no reports of anti-PD-1 neoadjuvant therapy for the dMMR/MSI-H colorectal cancer. Therefore, the aim of this study was to find the best multidisciplinary treatment for resectable colorectal cancer patient with the dMMR/MSI-H phenotype and to explore whether cyclooxygenase (COX) inhibitors combined with anti-PD-1 monoclonal antibody (mAb) could further improve efficacy.

DETAILED DESCRIPTION:
The PICC trial is an investigator-initiated, multi-cohort platform trial designed to evaluate the efficacy and safety of neoadjuvant toripalimab, with or without celecoxib, in patients with mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) locally advanced colorectal cancer. Each cohort within the PICC platform was independently conducted and analyzed according to prespecified objectives.

The initial exploratory cohort, PICC-1, was originally planned to enroll 20 eligible patients to receive neoadjuvant toripalimab plus celecoxib or toripalimab alone, with the primary objective of assessing feasibility and safety. The study was amended in August 2020 to change the primary objective to evaluating whether 6 cycles of neoadjuvant toripalimab with or without celecoxib improves the pathological complete response (pCR) rate compared with historical controls, with an updated planned enrollment of 34 eligible patients, who were to be randomized 1:1 between the two treatment groups. In May 2021, an additional 16 eligible patients were included in this exploratory cohort for translational research purposes.

The study was amended in April 2022 to add a new cohort, PICC-2, which was designed to formally compare the efficacy and safety of 12 cycles of neoadjuvant toripalimab plus celecoxib versus toripalimab monotherapy in patients with dMMR or MSI-H locally advanced colorectal cancer. A total of 110 eligible patients are planned to be randomized 1:1 between the two treatment groups.

The study was amended in June 2025 to add a new cohort, PICC-3, which was designed to evaluate the 3-year event-free survival (EFS) of 12 cycles of toripalimab plus celecoxib administered as neoadjuvant or definitive therapy in patients with dMMR or MSI-H locally advanced colorectal cancer. Approximately 108 eligible patients are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum.
3. Tumor tissues were identified as mismatch repair-deficient (dMMR) by immunohistochemistry (IHC) method or microsatellite instability-high (MSI-H) by polymerase chain reaction (PCR).
4. Male or female subjects aged 18 to 75 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Determined CT or MRI scans (done within 14 days of registration) of the chest, abdomen and pelvis: locally advanced (cT3-4 or cN1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]).
7. Non complicated primary tumor (obstruction, perforation, bleeding).
8. No previous any systemic anticancer therapy for colorectal cancer disease.
9. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women
8. Lack of effective contraception.
9. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
10. With any distant metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates (PICC-1 and PICC-2 cohorts) | 1 year
  The proportion of patients who achieved a pCR, which was defined as the absence of residual viable tumor cells in the primary tumor and all sampled lymph nodes at surgery.
Event-free survival (EFS) (PICC-3 cohort) | 3 years
  Defined as the time from randomization until the date of one of the following events (whichever occurred first): disease progression that precluded surgery, local R2 resection, local recurrence after an R0/1 resection, distant metastases, a new primary colorectal cancer, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Defined as the time from randomization to death from any cause.
R0 resection rates | 1 years
  The proportion of patients achieved a complete resection with negative margin.
Surgical and perioperative treatment safety | 1 years
  Assessed by evaluation of treatment-related adverse events
Surgery feasibility | 30 days after surgery
  Any treatment-related delays in the planned surgery of no more than 28 days after the last preoperative toripalimab dose

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Cao W, Hu H, Li J, Wu Q, Shi L, Li B, Zhou J, Wang X, Chen J, Wang C, Wang H, Deng W, Huang Y, Deng Y. China special issue on gastrointestinal tumors-Radiological features of pathological complete response in mismatch repair deficient colorectal cancer after neoadjuvant PD-1 blockade: A post hoc analysis of the PICC phase II trial. Int J Cancer. 2023 Dec 1;153(11):1894-1903. doi: 10.1002/ijc.34647. Epub 2023 Jul 6. PMID 37409565
- [Derived] Hu H, Kang L, Zhang J, Wu Z, Wang H, Huang M, Lan P, Wu X, Wang C, Cao W, Hu J, Huang Y, Huang L, Wang H, Shi L, Cai Y, Shen C, Ling J, Xie X, Cai Y, He X, Dou R, Zhou J, Ma T, Zhang X, Luo S, Deng W, Ling L, Liu H, Deng Y. Neoadjuvant PD-1 blockade with toripalimab, with or without celecoxib, in mismatch repair-deficient or microsatellite instability-high, locally advanced, colorectal cancer (PICC): a single-centre, parallel-group, non-comparative, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):38-48. doi: 10.1016/S2468-1253(21)00348-4. Epub 2021 Oct 22. PMID 34688374
- [Derived] Wang D, Cabalag CS, Clemons NJ, DuBois RN. Cyclooxygenases and Prostaglandins in Tumor Immunology and Microenvironment of Gastrointestinal Cancer. Gastroenterology. 2021 Dec;161(6):1813-1829. doi: 10.1053/j.gastro.2021.09.059. Epub 2021 Oct 2. PMID 34606846